CLINICAL TRIAL: NCT03196726
Title: POSTNATAL DEPRESSION: Malaysia ASPIRE* Project PHASE 2
Brief Title: Behavioural Interventions for Postnatal Depression: a RCT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, NOOR ANI AHMAD, Public Health Specialist, Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRR-15-2404-26677
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Postnatal Depression
Keywords: cognitive-behavioral therapy
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Management of postnatal depression mothers at primary care clinics using Cognitive-behavioural therapy treatment by nurses as adjunct to management by Medical Officer in intervention arm, compared to management by Medical Officer alone in control arm.
Who Masked: Participant, Care Provider
Masking Description: Participants randomized by offering 2 opaque envelope to group them into either as control or intervention group.
  Medical officers were responsible in the management of all participants using standard Clinical Practice Guideline (CPG). Participants from intervention group will see Medical Officer first before being given CBT by nurse
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will be seen by Medical Officer and manage using standard management based on Clinical Practice Guideline for management of postnatal depression. After session with Medical Officer, participants will be seen by Nurse who additionally manage them using brief Cognitive Behavioral Therapy. Participants will be follow-up at weekly basis for 6 weeks.
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy; Behavioral: standard management based on Clinical Practice Guideline
- Control arm (Placebo Comparator): Participants will be seen by Medical Officer and manage using standard management based on Clinical Practice Guideline for management of postnatal depression. Participants will be follow-up at weekly basis for 6 weeks.
  Interventions: Behavioral: standard management based on Clinical Practice Guideline

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Therapy — Week 1: Understanding postnatal depression Week 2: Relaxation techniques and tips to reduce stress Week 3: Positive thinking style and Self-Esteem Week 4: Relationship with partner Week 5: Relationship with infant Week 6: Relapse prevention
  Arms: Intervention Arm
Behavioral: standard management based on Clinical Practice Guideline — Mild depression: behavioral therapy; moderate depression: behavioral therapy and consider anti-depressant if required

SUMMARY:
Randomized-controlled trial on the effectiveness of managing postnatal depression mothers at primary care clinics using Cognitive-behavioural therapy treatment by nurses as adjunct to management by Medical Officer as compared to Medical Officer alone

DETAILED DESCRIPTION:
This was a two-group double-blind randomized controlled trial (RCT) conducted in six primary care clinics at Klang Valley, with 27 subjects in each arms. All post-partum women at 4 to 24 weeks, registered at these clinics, were screened using self-administered Edinburgh Postnatal Depression Scale for symptoms of depression. Those who scored 12 or more and/or positive for question on suicidal behaviour, were interviewed by trained Research Assistants using Mini International Neuropsychiatric Interview, a diagnostic interview tool. Those with mild to moderate depression were invited to join this study, while severe depressed cases were referred to the Family Medicine Specialist for appropriate management. Consented eligible women were randomized into either control group; managed by Medical Officers alone, or intervention group; managed by both Medical Officers and trained nurses. Medical officers were given standard refresher course on Postnatal Depression management based on Clinical Practice Guideline while nurses were trained using brief cognitive-behavioural therapy (CBT) module, which consists of 6 modules for 6 weekly sessions. Depression level and its severity were assessed using self-administered Beck's Depression Index (BDI) and Automatic Thought Questionnaire (ATQ), at Baseline, Week 3 and Week 6.

ELIGIBILITY:
Inclusion Criteria:

* postpartum 4-24 weeks
* registered with selected primary care clinics
* Edinburgh Postnatal Depression score: 12 or more; and Mini diagnostic interview:

positive (mild to moderate depression)

* consented to participate

Exclusion Criteria:

* severe depression or psychosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women postpartum 4 to 24 weeks
Enrollment: 54 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
changes in depression level | at baseline (Week 0), week 3 and Week 6
  assess changes in Beck Depression Index (BDI) score

CONTACTS AND LOCATIONS:
Overall Officials: Tahir Aris, MD, Study Director — INSTITUTE FOR PUBLIC HEALTH
Locations (6):
- Malaysia (6):
  - Klinik Kesihatan Seksyen 7,, Shah Alam, Selangor
  - Klinik Kesihatan Kuala Lumpur, Kuala Lumpur, W.P. Kuala Lumpur
  - Klinik Kesihatan Sg Besi, Kuala Lumpur, WP Kuala Lumpur
  - Klinik Kesihatan Presint 11, Putrajaya, WP Putrajaya
  - Klinik Kesihatan Presint 9, Putrajaya, WP Putrajaya
  - Klinik Kesihatan Presint 18, Putrajaya, WP Putraya

IPD SHARING:
Plan to Share IPD: No
data sharing must be requested from Director General of Health Malaysia